CLINICAL TRIAL: NCT01267838
Title: Randomised Comparison of T-stenting Versus Culotte Technique for the Treatment of de Novo Coronary Bifurcation Lesion With Drug-eluting Stents.
Brief Title: Culotte Technique Versus TAP Stunting for the Treatment of de Novo Coronary Bifurcation Lesion With Drug-eluting Stents
Acronym: BBK2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Responsible Party: Principal Investigator, Dr. Miroslaw FERENC, MD, University Heart Center Freiburg - Bad Krozingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBK2 study
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease; Restenosis
Keywords: Coronary artery disease; Restenosis; Stent thrombosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T Stenting group (Active Comparator): PCI of bifurcation lesion with modified T Stenting.
  Interventions: Procedure: PCI
- Culotte stenting group (Active Comparator): PCI of bifurcation lesion with Culotte stenting
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — PCI of bifurcation lesions with double stenting

SUMMARY:
BBK- 2 - study:

STUDY-SUMMARY

Background:

The need for stenting of the main and side branch (double stenting) in the treatment of coronary bifurcation lesion primarily depends on the complexity of the bifurcation lesion. If the bifurcation lesion is very complex (Medina classification 111, severe stenosis of both branches, severe calcified lesion, long lesions etc.) double stenting may be the treatment of choice. When double stenting is required, the most frequently used stenting techniques are T-stenting and Culotte-stenting. It is still unclear, however, which double stent technique yields the best long-term outcome.

Aim:

This randomized study will compare the long-term safety and efficacy of T-stenting versus Culotte-stenting in the treatment of de-novo coronary bifurcation lesions with drug-eluting stents.

Methods:

Three-hundred patients in whom a double-stenting technique is intended for the treatment of a de-novo coronary bifurcation lesion will be randomly assigned to T-stenting or Culotte-stenting with an approved drug-eluting stent. Patients will undergo 9-month angiographic follow-up with quantitative coronary angiography. Clinical follow-up is planed at 30 days, 6 months, 1 year, 2 years, 3 years and 5 years. The primary study endpoint is the maximal percent diameter stenosis in the bifurcation lesion at 9 months. Secondary endpoints include binary restenosis (estimated by Quantitative Coronary Angiography (QCA) analysis), Target Lesion Revascularisation (TLR), Freedom from Major Adverse Cardiac Events (MACE) and the rate of stent thrombosis according to the definition of the Academic Research Consortium (ARC definition). The study will have 90% power to detect a 25% reduction in the primary endpoint at p < 0.05.

DETAILED DESCRIPTION:
1. STUDY BACKGROUND:

Currently, a simple stepwise provisional T-stenting approach is most frequently used type of treatment in coronary bifurcation lesions. When stenting of both the side branch and the main branch (double stenting) is needed because of dissection, TIMI flow < 2, high residual stenosis > 75% there is a variety of techniques, which have been proposed. The most common techniques are T-stenting and Culotte-stenting.

Adriaenssens et al (1) have analysed the data of 132 patients treated with Culotte-stenting including Quantitative Coronary Angiography (QCA) analysis and clinical follow-up 1 year post Percutaneous Coronary Intervention (PCI). The authors demonstrated an incidence of binary angiographic restenosis of 22% for the whole bifurcation lesion. Procedural angiographic success was achieved in all lesions (final kissing balloon dilatation was performed in 62 % of patients). At 12 months, 28 of 132 (21%) patients had undergone target lesion revascularization. The incidence of stent thrombosis (at 1 year) was low (1.5%).

Ferenc et al. (2) compared systematic T-stenting with the provisional T-stenting in 202 patients of the BBK 1 study. There was no significant difference between the 2 strategies. Overall, maximum percent diameter stenosis in the bifurcation was 31 % at 9 months, corresponding to a binary restenosis rate of 11 %. Within 1-year follow-up, this prompted target lesion reintervention in 9,9 % of the patients. The risk of late stent thrombosis was low (2 %) at 2-year follow-up.

The randomised multicenter Nordic 2 study addressed the question whether Crush-stenting or Culotte-stenting achieves better angiographic and clinical outcome after PCI in bifurcation lesions (Erglis et al). The results demonstrated the superiority of Culotte-stenting as compared to the Crush-stenting. Major adverse cardiac events (MACE) as primary study endpoint occurred in 3.7 % in the Culotte study arm as compared to 4.3 in the Crush study arm (p =0.87). Likewise, in the double stent study arm of the BBC One study the Crush-stenting was used successfully (Hildick-Smith, TCT Late Breaking Trials 2008).

Currently, there is no data from randomized trials comparing T-stenting with Culotte-stenting.

References:

1. Adriaenssens, T., R. A. Byrne, et al: "Culotte stenting technique in coronary bifurcation disease: angiographic follow-up using quantitative coronary angiographic analysis and 12-months clinical outcomes." Eur Heart J 2008 29(23): 2868-76.
2. Ferenc M, Gick M, Kienzle RP, Bestehorn HP, Werner KD, Comberg T, et al. Randomized trial on routine vs. provisional T-stenting in the treatment of de novo coronary bifurcation lesions. Eur Heart J 2008;29(23):2859-67.
3. Erglis A, Kumsars I, Niemela¨ M, Kervinen K, Maeng M, Lassen JF, Gunnes P, Stavnes S, Jensen JS, Galløe A, Narbute I, Sondore D, Ma¨kikallio T, Ylitalo K, Christiansen EH, Ravkilde J, Steigen TK, Mannsverk J, Thayssen P, Nørregaard Hansen K, Syva¨nne M, Helqvist S, Kjell N, Wiseth R, Aarøe J, Puhakka M, Thuesen L; for the Nordic PCI Study Group. Randomized comparison of coronary bifurcation stenting with the crush versus the culotte technique using sirolimus eluting stents. Circ Cardiovasc Intervent. 2009;2: 27-34.
4. Hildick-Smith D, de Belder A, Cooter N et al. BBC ONE: The British Bifurcation Coronary study, Old New and Evolving strategies; a randomised trial of simple versus complex drug eluting stenting. TCT session -Late Breaking Trials 2008.

Trial randomisation scheme:

Time and Event Schedule

Event Screening Procedure 8-16-24 Hours 30 days 9 months 1 year 3 years 5 years Informed consent signed X Inclusion/Exclusion criteria X Medical History X X X X X X Angina pectoris status X X X X X X Creatine kinase (CK) and Troponin X X Medication History X X X X X X X Adverse Event Monitoring X X X X X X X (PCI) X Re - Angiography X

2. STUDY DESIGN

This study is a prospective, randomized, single-center evaluation of the treatment in de novo bifurcated coronary lesions comparing a technique of T-stenting with Culotte-stenting using approved drug- eluting stents.

The primary objective of this study is a comparison of T-stenting with Culotte-stenting with respect to the maximal percent diameter stenosis within the bifurcation at 9 months. In addition the study will assess various safety parameters.

Three-hundred patients will be enrolled in the study at one investigational site and will be randomly assigned to T-stenting or to Culotte-stenting of the bifurcation lesion. Any approved drug-eluting stent can be used. The choice of stent is left to the operator's discretion.

2.1 HYPOTHESIS

The hypothesis of this study is as follows:

In large coronary bifurcation lesions (main vessel ≥2.5mm, side branch ≥2.25mm) including significant ostial side branch disease, Culotte-stenting compared with T-stenting reduces maximal percent diameter stenosis at the bifurcation at 9-month follow-upby 25 %, relative. results in a lower restenosis rate than T stenting technique with a comparable long-term safety.

3. STUDY ENDPOINTS

3.1. Primary Study Endpoint

The primary study endpoint is:

- Maximal percent diameter stenosis at the bifurcation at 9 months.

3.2. Secondary Endpoints

The following secondary endpoints will be evaluated in this study:

* Binary restenosis (≥ 50% diameter stenosis) rate at any segment of the bifurcation at 9 month post procedure
* TLR of the main and side branch at 12 months post procedure.
* Binary restenosis (≥ 50% diameter stenosis) in the main and side branch at 9 months post procedure.
* MACE defined as death, Myocardial infarction (Q wave and Non-Q wave), emergent cardiac bypass surgery, or TLR at 30 days, 6 months, 1, 2, 3, 5 years.
* Device success defined as attainment of < 30% residual stenosis of the target lesion using drug-eluting stent (DES)in the main and side branch
* Procedure time, radiation time and volume of used contrast medium

  * Post-procedure thrombotic stent occlusion at 12 and 24 months according to the Academic Research Consortium-criteria:

Stent thrombosis is classified by the ARC definition as definite, probable, or possible and as early (0 to 30 days), late (31 to 360 days), or very late (>360 days).

The definition of definite stent thrombosis requires the presence of an acute coronary syndrome with angiographic or autopsy evidence of thrombus or occlusion.

Probable stent thrombosis includes unexplained deaths within 30 days after the procedure or acute myocardial infarction involving the target-vessel territory without angiographic confirmation.

Possible stent thrombosis includes all unexplained deaths occurring at least 30 days after the procedure. Intervening target-lesion revascularization is defined as any repeated percutaneous revascularization of the stented segment, including the 5-mm proximal and distal margins, that preceded stent thrombosis.

4 PATIENT SELECTION

This trial will include 300 patients with symptomatic de novo bifurcation lesion of a native coronary artery who meet eligibility criteria and agree to participate in the study.

4.1. Inclusion Criteria

Study candidates will be included only if all the following conditions are met:

1. Clinical indication for interventional treatment of the bifurcation lesion.
2. There is indication to perform the double stenting as judged by the operator.
3. Bifurcation lesions according to the Medina classification of a native coronary artery with a reference vessel diameter: main branch >2,5 mm; side branch >2,25 mm (the difference between vessel diameter of the main and side branch should be ≤1 mm)

   .
4. The target lesion (main branch and / or side branch) must be at least 50% diameter stenosis.
5. The target lesion has not been previously treated with any interventional procedure.
6. The target vessel (main branch and side branch) must be feasible for stent implantation (successful passage with the guide wire; successful predilatation with an appropriately sized balloon; no heavy calcification; no diffuse distal disease that might impede run off).
7. Patient has no other treatment planned within 30 days of the procedure.
8. Patient has been informed of the nature of the study and agrees to its provisions and has written informed consent as approved by the Ethics Committee.
9. Patient is willing to comply all required post-procedure follow-up.

4.2. Exclusion Criteria

Candidates will be excluded from participation in this study if any of the following conditions apply:

1. Patient had an acute myocardial infarction (> 3x normal CK ) within 72 hours preceding the index procedure and CK has not returned to normal limits at the time of the procedure.
2. Patient will have a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, prasugrel, stainless steel, sirolimus, everolimus, zotarolimus, biolimus or contrast sensitivity that cannot be adequately pre- medicated.
3. Non successful treatment of other lesion during the same procedure
4. Patient has a platelet count of <100,000 cells/mm³ or >700,000 cells/mm³, a White Blood Cells of <3,000 cells/mm³, or documented or liver disease.
5. Patient has a history of bleeding diathesis or coagulopathy.
6. Patient has suffered a stroke within the past six months.
7. Active peptic ulcer or upper gastrointestinal bleeding within the prior 6 months.
8. Patient has a co-morbidity (i.e. cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, or is associated with limited life- expectancy (less than 2 years).
9. Indication for oral anticoagulation
10. Patient must be excluded from the study if any of these angiographic criteria are met:

    1. The target vessel contains intraluminal thrombus.
    2. The target lesion or vessel shows angiographic evidence of severe calcification.
    3. The patient has undergone previous PCI to the target vessel within 6 months.
    4. Pre treatment of the lesion is done with a technique other than balloon angioplasty.

4.3 Randomisation

Patients who fulfil inclusion and exclusion criteria and give written informed consent to the study will be randomised according to a standard random number generation method. The study is designed as a non-blinded, randomized, single-center trial. Patients will be allocated to T-stenting or to Culotte-stenting using a computer-generated random sequence, set in blocks of 20 stratified to the type of drug-eluting stent in clinical use. The size of the block and the random sequence will be select by the statistician and will be unknown to the investigators and medical staff caring for the patients. Randomization will be performed immediately before catheter treatment of the bifurcation lesion.

5. PROCEDURES BY VISIT

5.1. Patient Enrollment

All potential subjects should be consented prior to performing any study related procedures. The investigator or representative will explain the nature and scope of the study, potential risks and benefits of participation, and answer questions for the patient and/or legally authorized representative. If the patient agrees to participate, the informed consent must be signed and dated; a copy must be provided to the patient or legally authorized representative.

Baseline data to be collected will include demographics , angiograophic and clinical parameters.

5.2. Laboratory Assessments

* ECG prior to procedure and between 12 hours and 24 hours post-procedure or before hospital discharge
* CK and CKMB and Troponin T prior to procedure and 8 hours, 16 hours and 24 hours post-procedure

5.3. Concomitant Medications

All subjects receive the medication regimen listed below. All medications administered should be recorded in the subjects medical record.

Prior to Procedure Aspirin At least 400 mg per os Clopidogrel 600 mg loading dose or Prasugrel 60 mg loading dose

During Procedure IV Heparin For angioplasty bolus 100 I.U./ kg/ KG IC Nitroglycerin 100 - 200 mcg prior to baseline and post intervention angiograms

Post-Procedure Aspirin At least 100 mg per day indefinitely Clopidogrel 75 mg per day for at least 6 months or Prasugrel 10 mg or 5 mg/die for at least 6 months as per clinical indication

Glycoprotein IIb/IIIa inhibitors (Abciximab) can be used only for bail out.

5.4. Coronary Angiography and Intervention

5.4.1. Angiography

Using standard procedures for angioplasty, an introducer sheath of at least 6 French will be introduced and the heparin bolus will be administered. After introduction of the guiding catheter and following intra-coronary injection of nitroglycerin, baseline angiography of the vessel will be performed in at least two best views that show the target lesion free of foreshortening or vessel overlap, using a 6 French or larger guiding catheter.

5.4.2. Lesion / Vessel Pre-treatment

For any patients with multiple lesions requiring treatment at the time of the index procedure, lesions outside the target vessel must be treated first successfully.

The target lesion in the main branch will be crossed with an intracoronary guide wire of 0.014 inch diameter and a second guide wire is passed into the side branch to protect the access. The choice of the appropriate guide wires is up to the discretion of the operator. After successful passage with the guide wires the lesion in the main branch should be pre-dilated with an appropriately sized balloon. Predilatation of the side branch before stenting of the main branch is up to the discretion of the operator.

5.4.3. Stenting Procedure and Stenting Technique

Among the many approaches to bifurcation stenting, we chose techniques that avoid non-stented gaps at the orifice of the side branch with minimal stent distortion or stent overlap in the carina region or the proximal segment of the main branch. Both techniques the provisional T-stenting as well the Culotte-stenting provide complete coverage of the side branch ostium. Final 'kissing balloon' dilatation should be performed in all patients irrespective of whether they were assigned to T-stenting or Culotte-stenting.

Stents should be selected long enough to cover the lesions completely. If more than one stent is needed to cover the lesion in the main or side branch completely, it is recommended to overlap the stents 1 - 2 mm. The aim should be to reach a diameter stenosis < 10% without proximal and distal dissections. Post dilatation may be performed at the operators discretion. Pre or post dilatation technique should avoid balloon injury to any segment of the vessel that will not be entirely covered by the drug eluting stent including the patients with provisional side branch stenting following an unsatisfactory result after balloon angioplasty.

T-stenting:

Both vessels have to be wired. Lesion preparation in the main vessel and side branch may be undertaken according to operator preference. After lesion preparation, the main branch is stented first.

After placement of the stent in the main branch, rewiring and predilatation of the side branch, the second stent in the side branch is advanced and an additional balloon is placed in the main branch at the orifice of the side branch. Then, the stent in the side branch is positioned, taking care that the marker band and about the first half millimetre of the stent are within the main branch stent. When the optimal position of the side-branch stent is achieved, the side-branch stent is deployedby a kissing balloon manoeuvre, first inflating the side-branch balloon with the stent and immediately afterwards the main branch balloon.

Culotte stent technique:

Both vessels have to be wired. Lesion preparation in the main vessel and side branch may be undertaken according to operator preference. After lesion preparation, the side branch have be stented first.

The first stent is placed from main branch into the side branch side branch, covering the entire diseased segment with a wire jailed in the main vessel. The main vessel is rewired through the stent struts, and after removal of the jailed wire, is dilated with a balloon to separate stent struts. The side branch wire is then removed (to prevent metal-to-metal jail) and the main vessel is stented covering the proximal and distal segment. The side-branch is re-wired and high pressure (e.g. 20 atm) individual inflations are made in each vessel at the bifurcation point to ensure good stent strut separation. Finally a lower pressure kissing inflation is made. For both the high pressure individual and lower pressure final kissing inflations, balloon sizing should be in accordance with the diameter of the vessel itself.

Further treatment to proximal or distal aspects of the main vessel or side branch can be continued at the discretion of the operator. At any stage, proximal or distal dissections may be treated as required with further stent implantations. At any stage, post-dilatations may be undertaken to optimise stent expansion.

Irrespective of the assigned treatment, glyceryl trinitrate is injected intra-coronarily at the completion of the procedure and final angiography of the vessel is performed in the two optimal views that were chosen at baseline.

5.4.4. Stent type

Any approved type of drug-eluting stent can be used at the operator's discretion.

5.5. Follow-up Procedures

All patients enrolled in the study will be required to complete 30 days, 6 months, one, two, three and fiv -years follow-up to evaluate long-term results.

5.5.1. 30 Days (± 5 days) Post Procedure (Telephone contact)

The assessment will include angina status (according to the Canadian Cardiovascular Society Classification of angina), all adverse events, all concomitant medications and any interventional treatment that occurred since the the index procedure.

5.5.2. Angiographic Follow-Up 9 Months (± 14 days) Post Procedure

As part of current routine clinical practice, all patients will undergo repeat angiography at 9 months after the index procedure. Angiographies will be performed as described in Section 5.4.1.

All films, including unscheduled angiograms, will be analysed to the angiographic core laboratory.

. 5.5.3. At 30 days, 6,12, 24. 36 and 60 Months (± 30 days) post Procedure (Telephone contact or contact with family doctor)

The assessment will include angina, all adverse events, all concomitant medications and any interventional treatment that occurred since the previous contact.

5.5.4 Quantitave coronary angiography:

For quantitative coronary angiography, angiograms obtained at baseline, at completion of the intervention and at 9 month follow-up will be analysed with using a computer based system dedicated to bifurcation analysis (Qangio XA, version7.0, Medis, Leiden, Netherlands), according to the standard operating procedure of our angiographic core laboratory. Quantitative angiographic measurements will be obtained of the three segments of the bifurcation lesion: the proximal and distal segment of the main branch and the side branch. We will perform measurements in the stented portion of the vessel (in-stent) and in the distal or proximal 5 mm margin (edge). In-segment analyses will comprise the in-stent and the edge area.

In addition, the bifurcation angle from the analysis system will be estimated.

6. SAFETY ISSUES

All serious adverse events must be reported to the ethic committee.

These include any complication that:

results in death is life-threatening results in persistent and significant disability or incapacity.

7. SAMPLE SIZE ESTIMATION

The study is designed to have a 90% power to detect a 25% relative reduction of the primary endpoint by Culotte technique as compared with T stenting at a significance level of 0.05. Assuming percent diameter stenosis in the side branch of 30±23 % at follow-up (ref. 10), a sample size of 133 patients in each arm is obtained. The study will include 150 patients in each arm, to allow for losses to angiographic follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for interventional treatment of the bifurcation lesion.
2. There is indication to perform the double stenting as judged by the operator.
3. Bifurcation lesions according to the Medina classification of a native coronary artery with a reference vessel diameter: main branch >2,5 mm; side branch >2,25 mm (the difference between vessel diameter of the main and side branch should be ≤1 mm)

   .
4. The target lesion (main branch and / or side branch) must be at least 50% diameter stenosis.
5. The target lesion has not been previously treated with any interventional procedure.
6. The target vessel (main branch and side branch) must be feasible for stent implantation (successful passage with the guide wire; successful predilataion with an appropriately sized balloon; no heavy calcification; no diffuse distal disease that might impede run off).
7. Patient has no other treatment planned within 30 days of the procedure.
8. Patient has been informed of the nature of the study and agrees to its provisions and has written informed consent as approved by the Ethics Committee.
9. Patient is willing to comply all required post-procedure follow-up.

Exclusion Criteria:

1. Patient had an acute myocardial infarction (> 3x normal CK ) within 72 hours preceding the index procedure and CK has not returned to normal limits at the time of the procedure.
2. Patient will have a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, prasugrel, stainless steel, sirolimus, everolimus, zotarolimus, biolimus or contrast sensitivity that cannot be adequately pre- medicated.
3. Non successful treatment of other lesion during the same procedure
4. Patient has a platelet count of <100,000 cells/mm³ or >700,000 cells/mm³, a White Blood Cells of <3,000 cells/mm³, or documented or liver disease.
5. Patient has a history of bleeding diathesis or coagulopathy.
6. Patient has suffered a stroke within the past six months.
7. Active peptic ulcer or upper gastrointestinal bleeding within the prior 6 months.
8. Patient has a co-morbidity (i.e. cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, or is associated with limited life- expectancy (less than 2 years).
9. Indication for oral anticoagulation
10. Patient must be excluded from the study if any of these angiographic criteria are met:

    1. The target vessel contains intraluminal thrombus.
    2. The target lesion or vessel shows angiographic evidence of severe calcification.
    3. The patient has undergone previous PCI to the target vessel within 6 months.
    4. Pre treatment of the lesion is done with a technique other than balloon angioplasty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-02; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximal percent diameter stenosis at the bifurcation (QCA) | 9 months post index PCI
  Maximal percent diameter stenosis at the bifurcation (QCA)

SECONDARY OUTCOMES:
TLR of the main and side branch | 12 months post index PCI
  TLR of the main and side branch at 12 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw Ferenc, MD, Principal Investigator — Herz-Zentrum Bad Krozingen
Locations (1):
- Herz-Zentrum Bad Krozingen, Bad Krozingen, Suedring 15, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferenc M, Gick M, Kienzle RP, Bestehorn HP, Werner KD, Comberg T, Kuebler P, Buttner HJ, Neumann FJ. Randomized trial on routine vs. provisional T-stenting in the treatment of de novo coronary bifurcation lesions. Eur Heart J. 2008 Dec;29(23):2859-67. doi: 10.1093/eurheartj/ehn455. Epub 2008 Oct 9. PMID 18845665
- [Background] Adriaenssens T, Byrne RA, Dibra A, Iijima R, Mehilli J, Bruskina O, Schomig A, Kastrati A. Culotte stenting technique in coronary bifurcation disease: angiographic follow-up using dedicated quantitative coronary angiographic analysis and 12-month clinical outcomes. Eur Heart J. 2008 Dec;29(23):2868-76. doi: 10.1093/eurheartj/ehn512. Epub 2008 Nov 11. PMID 19001472
- [Background] Erglis A, Kumsars I, Niemela M, Kervinen K, Maeng M, Lassen JF, Gunnes P, Stavnes S, Jensen JS, Galloe A, Narbute I, Sondore D, Makikallio T, Ylitalo K, Christiansen EH, Ravkilde J, Steigen TK, Mannsverk J, Thayssen P, Hansen KN, Syvanne M, Helqvist S, Kjell N, Wiseth R, Aaroe J, Puhakka M, Thuesen L; Nordic PCI Study Group. Randomized comparison of coronary bifurcation stenting with the crush versus the culotte technique using sirolimus eluting stents: the Nordic stent technique study. Circ Cardiovasc Interv. 2009 Feb;2(1):27-34. doi: 10.1161/CIRCINTERVENTIONS.108.804658. Epub 2009 Feb 10. PMID 20031690
- [Background] Hildick-Smith D, de Belder AJ, Cooter N, Curzen NP, Clayton TC, Oldroyd KG, Bennett L, Holmberg S, Cotton JM, Glennon PE, Thomas MR, Maccarthy PA, Baumbach A, Mulvihill NT, Henderson RA, Redwood SR, Starkey IR, Stables RH. Randomized trial of simple versus complex drug-eluting stenting for bifurcation lesions: the British Bifurcation Coronary Study: old, new, and evolving strategies. Circulation. 2010 Mar 16;121(10):1235-43. doi: 10.1161/CIRCULATIONAHA.109.888297. Epub 2010 Mar 1. PMID 20194880